CLINICAL TRIAL: NCT03010189
Title: Actigraphy and Nocturnal Heartrate Variability in Cluster Headache Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordlandssykehuset HF (Other)
Collaborators: University of Tromso (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/1789(REK)
Record Dates: First submitted 2016-07-27; First posted 2017-01-04 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Cluster Headache; Sleep
Keywords: Cluster headache; Actigraphy; Pupillometry
MeSH Terms: conditions — Cluster Headache | interventions — Actigraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patient (Experimental): Cluster headache patients are examined with light reflex pupillometry, two weeks actigraphy and heart-rate variability monitoring both in headache phase and remission phase.
  Interventions: Device: Actigraphy; Device: Heart-rate variability monitoring; Device: Pupillometry
- Controls (Active Comparator): Healthy controls undergo the same examinations once: light reflex pupillometry, actigraphy and heart-rate variability monitoring.
  Interventions: Device: Actigraphy; Device: Heart-rate variability monitoring; Device: Pupillometry

INTERVENTIONS:
Device: Actigraphy — A small computer in the shape of a wristwatch, that registers movement and assesses sleep quality.
Device: Heart-rate variability monitoring — A small computer that registers variation in heart rate, which reflects cardiac autonomic tone.
Device: Pupillometry — A handheld infrared camera that sends out a light flash and records the pupil as it contracts and dilates, as a measure of pupillary autonomic tone.

SUMMARY:
Cluster headache is one of the most painful headaches, characterized by recurring episodes of unilateral, periorbital pain, which is accompanied by autonomic symptoms that seem to be of both sympathetic and parasympathetic origin. The pathophysiology behind the condition is largely unknown, but increasing evidence indicate that the hypothalamus plays a pivotal role. The headache attacks come in clusters or bouts (hence the name) which last up to three months, after which the headache disappears for at least one month. 10-15% have chronic cluster headache. During attacks, the patients have cranial sympathetic hypoactivity and parasympathetic hyperactivity, whereas they have cranial parasympathetic hypoactivity during remission phase. There is an emerging hypothesis that headache attacks are elicited in a state of autonomic hypoarousability, which is also supported by the fact that most cluster attacks occur during the night, when the patients are sleeping.

The aim in this project is to study the intercept between the sleep-wake cycle, autonomic tone and the occurrence of headache attacks, by using actigraphy, heart-rate variability and pupillometry. All these methods are well validated, and frequently used in studies on sleep and autonomic function. The study design is that of a case-control model where 15 cluster headache patients will undergo pupillometry, before wearing the actigraph and heart-rate variability-monitor for two weeks, once in cluster bout and once in remission phase. The actigraphy will register nocturnal movement and sleep quality, and headache attacks will be registered by pressing a button on the actigraph. The pupillometry measures pupillary constriction and dilation in response to light, a reflex that is controlled by the autonomic nervous system. The heart-rate variability monitors fluctuations in the heart rate which reflects the sympathovagal balance of cardiac control. All participants will fill out the Pittsburgh Sleep Quality Index before and after registration. In addition, 15 healthy controls will undergo one session of the same examinations. The results of the study will give valuable insight to the pathophysiology of a condition that is very painful and has great impact on the patients' quality of life, and also add knowledge to the relation between headache, sleep and the autonomic nervous system.

DETAILED DESCRIPTION:
Cluster headache (CH) is a primary headache in which recurring episodes of unilateral, periorbital pain is accompanied by unilateral autonomic symptoms such as tearing, conjunctival injection, nasal congestion or rhinorrhea, miosis and ptosis. Headache attacks last from 15 to 180 minutes, and patients may have up to eight attacks each day. Most attacks occur at night between midnight and 04 a.m. Headache attacks come in recurring bouts lasting up to three months, after which the headache disappears for at least one month. 10-15% of patients have chronic cluster headache, meaning that there are no pauses between bouts. The condition has a prevalence of about 0.2% and affects men 3-4 times more often than women.

The combination of unilateral headache and autonomic symptoms makes CH an interesting disorder to study in view of headache pathophysiology. Increasing amounts of evidence points at the hypothalamus as the locus in quo for CH pathophysiology. During attacks, the autonomic symptoms seem to be caused both by a hypofunction of sympathetic activity (miosis and ptosis), and a hyperfunction of parasympathetic activity (conjunctival injection, tearing and nasal congestion). Physiological studies seem to imply that patients during bouts have an upregulated parasympathetic activity caused by activation of the trigemino-parasympathetic reflex and a downregulated sympathetic tone, while they outside of bouts have a downregulated parasympathetic tone. Studying the autonomous nervous system in cluster headache patients is difficult, as they usually have headaches only a few months during the year and the attacks are quite short lasting, but excruciating painful when they occur, leaving the patients restless and with an urge to move about. This makes it difficult to study what actually happens during the painful phase. Thus, finding new ways to study the autonomic nervous system in these patients during the various stages of their disease is very important.

In addition to autonomic dysfunction, sleep disturbances are frequent and well documented in CH patients. Sleep is often problematic in all headaches, but CH patients seem to have a high prevalence of insomnia even when compared to other headache populations. This is not merely a result of the recurring nocturnal headaches, as CH patients have significantly reduced sleep quality compared to controls even one year after last headache attack. The documentation mostly consist of studies using well validated questionnaires such as the Pittsburgh Sleep Quality Index (PSQI) or diagnostic criteria such as the DSM IV. Only one major study have assessed sleep quality in cluster headache using quantitative methods such as polysomnography. In this study, the authors found that cluster headache patients in headache bout had a reduced percentage of REM sleep, longer REM latency and fewer arousals compared to healthy controls. There was no temporal relationship between headache attacks and specific sleep stages. Sleep is the single most important trigger for attacks in cluster headache, and most attacks occur during the late night or early morning hours.

We know that the balance between sympathetic and parasympathetic tone differ between REM and NREM-sleep stages in healthy individuals, and that there is a transient decrease in sympathetic tone during the night, which is reflected in a period of reduced heart rate and blood pressure. This "dipping" coincides with the increased occurrence of cluster attacks, and fits well into the emerging theory that cluster headache attacks is elicited in a state of hypoarousability, or reduced sympathetic tone. Thus, sleep disturbances are, together with autonomic dysfunction, an integral part of CH pathophysiology, and further studies are needed to elucidate the association between sleep, autonomic dysfunction and headache attacks.

The aim of this study is to assess sleep quality and autonomic tone in CH patients inside and outside of headache bouts, compared to healthy controls. Inside of bouts, the investigators will assess how the occurrence of headache attacks are related to autonomic tone. The data will be gathered by using actigraphy, pupillometry and heart-rate variability, all well validated research tools. In addition, all participators will fill out the PSQI reporting subjective sleep quality.

Pupillometry: The pupillary response to light is conducted by the autonomous nervous system. In short, constriction of the pupil is a parasympathetic response, and pupillary redilation a sympathetic response. By measuring the velocity of constricting and dilating the pupil, you get a good view of the balance between the two. The measurements are made in 1 lux ambient darkness with a pupillometer that consists of a infra-red camera that films the pupil as it responds to a small light flash, and measures the time the pupil takes to contract and redilate again.

Heart-rate variability: Heart-rate variability (HRV) is an indirect, non-invasive way of measuring the autonomic nervous system activity, with contributions from both the sympathetic and parasympathetic nervous systems. Frequency-specific fluctuations in the heart rate are assessed with power spectrum analysis. The high frequency component (HF: 0.15-0.4 Hz) reflects vagal control, whereas the low frequency component (LF: 0.04-0.15) reflects sympathetic control. The LF/HF ratio reflects sympathovagal balance. Reduced Heart-rate variability has been associated to increased mortality in patients with myocardial infarction and heart failure. A simple computer placed on the forearm combined with a monitor placed on the chest, giving minimal discomfort to the patient, may now measure heart rate variability.

Actigraphy: Polysomnography is the gold standard of sleep assessment, but is quite an extensive and resource intensive method. In later years, new technology has made actigraphy a reliable and easy way to measure sleep in a less invasive manner. An actigraph is a small, wrist-watch-sized device that monitors movement by using an accelerometer that tracks motion and creates a graph. In addition, a button can be pushed to mark events such as bedtime or waketime. Actigraphs are widely used to study sleep-wake cycles and circadian rhythms. Several studies have compared actigraphy to polysomnography in the assessment of e.g. insomnia and other sleep disturbances, and found it to be a valid and cost-effective alternative.

The Pittsburgh Sleep Quality Index: There are several self-report questionnaires available measuring subjective sleep quality, and the Pittsburgh sleep quality index is one of the best validated and widely used alternatives. PSQI measures retrospective subjective sleep quality and disturbances during the last month.

The study will be conducted as a case-control study, comparing patients to healthy controls, but it will also compare patients to themselves in and out of headache bouts. The patients will undergo pupillometry, actigraphy and HRV registration twice: once in remission phase, and once in headache phase. Pupillometry will be conducted at the out-patient clinic. Here, the participants will also receive their actigraph and HRV-monitor. Each registration will last two weeks, where the actigraph, formed as a watch, is placed on the patient's wrist for recording of movement during day and night, and a heart rate monitor formed as a belt records heart rate variability. Software is available to interpret the data making it possible to measure sleep and vasoactive tone. After the two weeks are over, the patients will fill out the PSQI, reporting the subjective sleep quality, which may be compared to the registrations from the actigraph. To register in headache phase, the patients must be willing to contact the study researchers and give notice when the bout has begun, so that they may come and receive the actigraph. The patients will be asked to mark the occurrence of attacks during the registration by pressing a button on the actigraph.

The healthy controls will undergo pupillometry, actigraphy and HRV monitoring only once, and fill out the PSQI after registration. The PSQI also registers the use of sleeping pills, which may be used in both patients and controls. For each two weeks registration, the average number of hours with daylight will be noted, as this may influence the sleep quality of the patients. These data will be given from the Norwegian Meteorological Institute.

ELIGIBILITY:
Inclusion Criteria:

* Episodic or chronic cluster headache, according to the ICHD-IIIb criteria.

Exclusion Criteria:

* Cardiac arrythmia or known autonomic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in pupillary average contraction velocity | Once in the beginning of a headache phase, and once 4 weeks after last headache attack
  The velocity of pupillary constriction in response to light, measured with a pupillometer, in mm/sec
Change in total sleep time | Measured for two weeks during headache phase, and again four weeks after last headache attack
  Average number of hours asleep per night, measured over two weeks with an actigraph
Change in sleep efficiency | Measured for two weeks during headache phase, and again four weeks after last headache attack
  Average number of hours asleep per night divided by time spent in bed, measured over two weeks with an actigraph
Change in wake after sleep onset | Measured for two weeks during headache phase, and again four weeks after last headache attack
  Average number of awakenings during the sleep phase, measured over two weeks with an actigraph
Change in LF/HF ratio | Measured for two weeks during headache phase, and again four weeks after last headache attack
  The ratio of low-frequency and high-frequency fluctuations in heart rate, measured over two weeks with a heart-rate variability monitor

CONTACTS AND LOCATIONS:
Overall Officials: Karl B Alstadhaug, MD, PhD, Principal Investigator — Nordlandssykehuset HF
Locations (1):
- Nordland Hospital Trust, Bodø, Nordland, Norway

IPD SHARING:
Plan to Share IPD: No